CLINICAL TRIAL: NCT05189847
Title: Clinical Register Studying the therApeutic Patient Population With Multifocal Atherosclerosis in the Russian Federation and Eurasian Countries
Brief Title: Clinical Register Studying the therApeutic Patient Population With Multifocal Atherosclerosis
Acronym: KAMMA
Status: Completed | Type: Observational
Sponsor: Eurasian Association of Therapists (Other)
Responsible Party: Sponsor
Other Study IDs: KAMMA
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Polyvascular Disease; Atherosclerosis; Atherosclerosis Generalized; Cardiovascular Diseases; Cardiac Death; Chronic Kidney Diseases; Bleeding; Acute Stroke; Acute Coronary Syndrome
Keywords: Atherosclerosis; polyvascular disease; cardiovascular diseases; acute stroke; acute coronary syndrome; cardiac death; Chronic kidney disease; bleeding; hospitalization; amputation; cardiovascular event; cerebrovascular accident
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Death; Renal Insufficiency, Chronic; Hemorrhage; Stroke; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with MFA: Patients with MFA confirmed by ultrasound examination, ABI or using clinical and medical history data.
- Patients with a history of established isolated coronary artery disease: The criterion for inclusion of patients in the present study is the diagnosed ischemic heart disease.

SUMMARY:
Аn international, multicenter, non-interventional real-life clinical practice Register studying the Actual therapeutic patient population with Multifocal Atherosclerosis in the Russian Federation and Eurasian countries

DETAILED DESCRIPTION:
Information on demographics, comorbidities, methods for diagnosing multifocal atherosclerosis (MFA), prescribed therapy, and outcomes will be identified via medical records analysis. Results of arterial bed ultrasound examination (US), results of ankle-brachial index (ABI) measurements, along with clinical and anamnestic data on target organ damage in the MFA-affected areas will be used as the main source verifying the presence MFA.

The follow-up period for each patient will span from the date of inclusion and over the next year with an additional 6 and 12 months of follow-up.

Patients eligible for entry in the Register must be included and their details must be documented. The procedure for obtaining informed consent for the examination and collection of data must comply with the requirements of local legislation. Patients will be required to sign an informed consent document if required.

Standardized electronic CRFs will be used in all research centers. The electronic data collection (EDC) system must be validated in accordance with current standards and legal requirements. Researchers will log into this system using individually assigned usernames and passwords. Data can only be entered and corrected by the researcher or other authorized personnel of the research center.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 and older at the time of data registration; Presence of 2 or more of the following factors

  * Coronary arteries atherosclerosis (atherosclerosis revealed by means of coronary angiography and/or a history of type I myocardial infarction and/or elective PCI and/or CABG and/or angina pectoris with ischemia according to stress test results, history of CHD);
  * Lower extremity arteries atherosclerosis (atherosclerotic plaques revealed by ultrasound, and/or ABI <0.9, and/or a history of revascularization, and/or a history of amputation associated due to chronic lower extremities arterial insufficiency);
  * Atherosclerosis of brachiocephalic arteries or renal arteries (presence of atherosclerotic plaques according to US data and/or history of revascularization and/or history of atherothrombotic stroke or TIA in the absence of known AF);
  * Atherosclerosis of renal arteries or abdominal aorta (presence of atherosclerotic plaques according to US data and/or history of revascularization).

Presence of one or more of the following atherosclerotic risk factors:

* Anamnestic data on dyslipidemia with LDL cholesterol levels above 4.9 mmol/L or total cholesterol levels above 8.0 mmol/L;
* Presence of confirmed familial hypercholesterolemia;
* Current smoker status or history of smoking;
* Overweight (BMI≥ 25 kg/m2);
* Presence of arterial hypertension;
* Presence of established type 2 diabetes mellitus;
* Presence of an established diagnosis of prediabetes;
* Presence of CKD stage 3a and higher (GFR <60 ml / min / 1.73 m2).

Exclusion Criteria:

* Life expectancy less than 1 year;
* Patient refusal to participate in the Register

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anonymized male and female patients over 18 years and suffering MFA confirmed by ultrasound method, ankle-brachial index along with clinical and anamnestic data.
Sampling Method: Probability Sample
Enrollment: 3059 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of a cardiovascular event (stroke, ACS, amputation, hospitalizations (related or not to cardiovascular pathology), the number of emergency calls) | after 12 months
  To assess the occurrence of cardiovascular events in 6 and 12 months in a cohort of patients with MFA: brain hemorrhage, acute coronary syndrome, amputation, admission to hospital (related or not related to a cardiovascular disease), number of emergency calls

SECONDARY OUTCOMES:
All-cause mortality | after 12 months
  To estimate overall mortality at 6 and 12 months in a cohort of patients with MFA
The frequency of any bleeding episodes (life-threatening, bothersome, or of unknown severity) | after 12 months
  To evaluate bleeding at 6 and 12 months in a cohort of patients with MFA
Change of GFR according to Chronic Kidney Disease Epidemiology Collaboration | after 12 months
  To compare the course of CKD in different subpopulations of patients
Prevalence of risk factors in the population | after 12 months
  To estimate the prevalence of risk factors in the population
Change of 3 point major adverse cardiovascular events parameter (Cardiovascular death, Nonfatal stroke, Non-fatal myocardial infarction) | after 12 months
  To evaluate patients according to 3P MACE parameter ((Cardiovascular death, Nonfatal stroke, Non-fatal myocardial infarction) according to prescribed therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Arutyunov, professor, Study Chair — Eurasian Association of Therapists
Locations (1):
- Eurasian Association of Therapists, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study design — http://doi.org/10.17802/2306-1278-2023-12-2-6-13
- See also: Peculiarities of polyvascular disease and the diagnostic significance of the ankle-brachial index in patients with coronary artery disease: results from the real-world registry KAMMA — http://doi.org/10.15829/1560-4071-2024-5837